CLINICAL TRIAL: NCT03207425
Title: A Phase 1, Open-Label, Parallel Group, Single Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of EDP 305 in Subjects With Varying Degrees of Hepatic Function
Brief Title: A Study of EDP-305 in Subjects With Mild and Moderate Hepatic Impairment Compared With Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 305-003
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-06

CONDITIONS: NASH
Keywords: Hepatic Impairment

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment group (Experimental)
  Interventions: Drug: EDP 305
- Moderate hepatic impairment group (Experimental)
  Interventions: Drug: EDP 305
- Matching healthy control group (Experimental): Healthy control group will be matched with the hepatically impaired population with respect to age, sex and BMI
  Interventions: Drug: EDP 305

INTERVENTIONS:
Drug: EDP 305 — Each subject will receive a single dose of EDP 305 on Day 1.

SUMMARY:
This is a study to characterize the pharmacokinetics as well as safety and tolerability of a single oral dose of EDP-305 in subjects with mild and moderate hepatic impairment compared to matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the ICF and able to comply with the study restrictions
* Adult male or female subjects age 18 to 75 years, inclusive, at the time of informed consent
* Female subjects must be non-childbearing potential

Additional criteria for hepatically impaired subjects

* Confirmed diagnosis of cirrhosis due to parenchymal liver disease
* Stable hepatic impairment, defined as no clinically significant change in disease status, as judged by the Investigator

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at Screening that the Investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer except for conditions associated with hepatic impairment in subjects with compromised hepatic function
* Clinically significant renal disease

Additional criteria for hepatically impaired Subjects

* History of esophageal bleeding within the last 3 months prior to study drug administration
* Severe hepatic encephalopathy (Grade >2) or degree of central nervous system (CNS) impairment
* History of liver transplantation
* Presence of Hepatocellular Carcinoma, or suspicion of Hepatocellular Carcinoma based on Investigator's judgment
* Hepato-renal or hepato-pulmonary syndrome
* Prior placement of a portosystemic shunt
* Spontaneous bacterial peritonitis currently or within the last 6 months
* Hospitalization within the last 2 months related to cirrhosis
* Advanced ascites and ascites which require emptying and albumin supplementation, as judged by the Investigator
* Hemoglobin concentration < 10.0 g/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP 305 | From pre-dose on Day 1 until 216 hour post-dose (Day 10)
AUCinf of EDP 305 | From pre-dose on Day 1 until 216 hour post-dose (Day 10)
t1/2 of EDP 305 | From pre-dose on Day 1 until 216 hour post-dose (Day 10)
CL/F of EDP 305 | From pre-dose on Day 1 until 216 hour post-dose (Day 10)

SECONDARY OUTCOMES:
Safety measured by adverse events, physical exams, vital signs, 12-lead electrocardiograms (ECGs) and clinical lab results (including chemistry, hematology, and urinalysis). | From Screening up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (3):
- American Research Corporation at The Texas Liver Institute, San Antonio, Texas, United States
- Pharmaceuticals Research Associates, Prague, Czechia
- Summit SRO, Bratislava, Slovakia